CLINICAL TRIAL: NCT03249740
Title: A Phase 1/2 Multicenter Study Evaluating the Safety, Tolerability, and Efficacy of an Intravitreal Depot Formulation of Sunitinib Malate (GB-102) in Subjects With Neovascular Age-related Macular Degeneration
Brief Title: A Depot Formulation of Sunitinib Malate (GB-102) in Subjects With Neovascular (Wet) Age-related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Graybug Vision (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GBV-102-001
Record Dates: First submitted 2017-08-02; First posted 2017-08-15 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: Age-related macular degeneration; Choroidal neovascularization
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Sunitinib; aflibercept

STUDY DESIGN:
Intervention Model Description: Phase 1: open-label GB-102 dose cohorts are initiated sequentially Phase 2: assignment to and initiation of cohorts occur in parallel - not completed in this study. Separate protocol (GBV-102-002) implemented for Phase 2.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Masking is relevant to Phase 2 only
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental: Phase 1 - GB-102 (Experimental): Subjects will be assigned to 1 of 4 cohorts to receive a single intravitreal injection of up to 2.0 mg (50 μL) GB-102.
  Interventions: Drug: GB-102
- Experimental: Phase 2 - GB-102 (Experimental): Low dose or high dose injected every 6 months
  Interventions: Drug: GB-102
- Active Comparator: Phase 2 - Aflibercept (Active Comparator): Aflibercept 2 mg injected every 2 months
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: GB-102 — Intravitreal injection of GB-102
  Other Names: Sunitinib malate
  Arms: Experimental: Phase 1 - GB-102; Experimental: Phase 2 - GB-102
Drug: Aflibercept — Intravitreal injection of Aflibercept.
  Other Names: Anti-VEGF
  Arms: Active Comparator: Phase 2 - Aflibercept

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of single and repeated intravitreal injections of GB-102 in subjects with neovascular (wet) age-related macular degeneration.

DETAILED DESCRIPTION:
In this 2-part study, Part 1 is a multicenter, open-label, safety, tolerability, and systemic exposure evaluation to Sunitinib in escalating doses of a single IVT injection of GB-102, while Part 2 is a multicenter, double-masked, randomized (1:1:1), parallel-group, safety, and efficacy evaluation of repeated IVT injections of 2 dose levels of GB-102 compared with aflibercept.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males or females of any race, ≥ 50 years of age
2. Presence of an active CNV lesion secondary to AMD treated with at least 3 monthly injections of an anti-VEGF agent (aflibercept, bevacizumab, or ranibizumab)
3. Evidence of increased vascular permeability and/or loss of visual acuity

Key Exclusion Criteria:

1. History, within 6 months prior to screening, of any of the following: myocardial infarction, any cardiac event requiring hospitalization, treatment for acute congestive heart failure, transient ischemic attack, or stroke
2. Uncontrolled hypertension, diabetes mellitus, IOP, hypothyroidism, or hyperthyroidism
3. Chronic renal disease
4. Abnormal liver function
5. Women who are pregnant or lactating

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
Phase 1: Occurrence of ocular and nonocular adverse events (AEs) | 8 months
  Number of adverse events in total and number of subjects with an adverse event
Phase 2: Change from baseline in best corrected visual acuity by ETDRS | Baseline, Month 9
  Mean change from Baseline at Day 270 (Month 9) in best corrected visual acuity (BCVA) measured by early treatment diabetic retinopathy (ETDRS)

SECONDARY OUTCOMES:
Phase 1: Change from baseline in BCVA by ETDRS | 8 months
  Mean change from baseline in mean BCVA measured by early treatment diabetic retinopathy (ETDRS) method
Phase 1: Change from baseline in sub-retinal thickness | 8 months
  Mean change from baseline in sub-retinal thickness (microns) by spectral domain - optical coherence tomography (SD-OCT)
Phase 1: Change from baseline in retinal fluid by SD-OCT | 8 months
  Assessment of retinal fluid by SD-OCT
Phase 1: Change from baseline in total lesion area by FA/CFP | 8 months
  Lesion area (total) by fluorescein angiography/color fundus photography (FA/CFP)
Phase 1: Change from baseline in CNV lesion area by FA/CFP | 8 months
  CNV lesion area by FA/CFP
Phase 1: Change from baseline in fluorescein leakage area by FA/CFP | 8 months
  Area of fluorescein leakage by FA/CFP
Phase 1: Rescue medication | 8 months
  Proportion of subjects receiving rescue medication and median time to rescue medication
Phase 1: Systemic exposure to sunitinib measured in plasma level | 8 months
  Plasma levels of sunitinib (ng/mL)
Phase 1: Change from baseline in sub retinal hyper reflective material (SHRM) height | 8 months
  Subretinal hyper reflective material (SHRM) height
Phase 2: Proportion of subjects with absence of retinal fluid by SD-OCT | 12 months
  Assessment of retinal fluid by SD-OCT
Phase 2: Proportion of subjects with < 15 BCVA letter loss by ETDRS | 12 months
  Proportion of subjects with < 15 letters lost in BCVA measured by ETDRS method, baseline comparison to assessments at months 1-12
Phase 2: Proportion of subjects with ≥ 15 BCVA letters gained by ETDRS | 12 months
  Proportion of subjects with ≥ 15 letters gained in BCVA measured by ETDRS method, baseline comparison to assessments at months 1-12
Phase 2: Occurrence of ocular and nonocular adverse events (AEs) | 12 months
  Number of adverse events in total and number of subjects with an adverse event
Phase 2: Change from baseline in BCVA by ETDRS | 12 months
  Mean change from baseline in mean BCVA measured by early treatment
Phase 2: Systemic exposure to sunitinib measured in plasma level | 12 months
  Plasma levels of sunitinib (ng/mL)
Phase 2: Change from baseline in sub-retinal thickness | 12 months
  Mean change from baseline in sub-retinal thickness (microns) by SD-OCT
Phase 2: Rescue medication | 12 months
  Proportion of subjects receiving rescue medication and median time to rescue medication

CONTACTS AND LOCATIONS:
Overall Officials: Charles P. Semba, MD, Study Director — Graybug Vision, Inc.
Locations (8):
- United States (8):
  - Retinal Consultants of Arizona, Gilbert, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Midwest Eye Institute, Indianapolis, Indiana
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Arlington, Texas
  - Retina Research Center, PLLC, Austin, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas